CLINICAL TRIAL: NCT01701830
Title: The Relationship Between Serum Omentin-1 and IL-6 and Carotid Atherosclerosis In Non-Diabetic Chronic Kidney Disease
Brief Title: Serum Omentin-1 and Carotid Atherosclerosis In Non-Diabetic Chronic Kidney Disease
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Kocaeli Derince Education and Research Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 2012/02
Record Dates: First submitted 2012-10-03; First posted 2012-10-05 (Estimated); Last update posted 2012-10-05 (Estimated); Status verified 2012-10

CONDITIONS: Non-diabetic Chronic Kidney Disease; Atherosclerosis
Keywords: omentin-1; carotid atherosclerosis; kidney disease
MeSH Terms: conditions — Atherosclerosis; Carotid Artery Diseases; Kidney Diseases

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional

GROUPS / COHORTS (2):
- Case Group: Patients with chronic kidney disease of stage 3-4.
- Control group: 30 healthy subject

SUMMARY:
The aim of the study is to evaluate whether a low level of serum omentin-1 is associated with carotid atherosclerosis and mediated by inflammation.

DETAILED DESCRIPTION:
Atherosclerotic cardiovascular disease is markedly increased in chronic kidney disease. There are a lot of risk factor, along with conventional risk factors. Serum onemtin-1 is a adipokine and suggested as a new marker for vascular disease.It has some anti-atherogenic properties. Studies investigating serum omentin-1 level have usually conducted in patients with diabetes mellitus.

ELIGIBILITY:
Inclusion Criteria:

* between ages of 18 - 65 years old chronic kidney disease of stage 3-4

Exclusion Criteria:

* Chronic kidney disease of stage 5
* The history of ischemic cardiovascular disease (myocardial infarction, unstable angina, stroke, peripheral artery disease, or cardiovascular revascularization)
* Severe heart failure
* Stage 2 hypertension
* Diabetes mellitus
* Corticosteroid therapy
* Severe hepatic disease
* Smoking
* Inflammatory disease
* Acute infectious disease
* Malignancy

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Department of Nephrology, Check-up clinic
Sampling Method: Non-Probability Sample
Enrollment: 85 (Estimated)
Dates: Start 2012-10; Study Completion 2013-05 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Erkan SENGUL, MD, Principal Investigator — Kocaeli Derince Education and Training Hospital
Locations (1):
- Department of Nephrology, Check-up Clinic,Kocaeli Derince Education and Traning Hospital, İzmit, Kocaeli, Turkey (Türkiye)